CLINICAL TRIAL: NCT02073045
Title: Effect of Intensive Education on Breast Cancer Patient's Understanding of Lymphedema
Brief Title: Intensive Education in Increasing Understanding of Lymphedema in Patients With Breast Cancer Undergoing Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: research cancelled
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1113; NCI-2014-00348 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 1113 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care (lymphedema education) (Experimental): In an educational intervention, participants complete a five question lymphedema survey, designed by the Occupational Therapy staff, as an instrument to assess a patient's knowledge of lymphedema signs/symptoms before surgery. An OT, PT, and/or CLT provide written handouts to participants on the pathophysiology, signs, symptoms, and treatment of lymphedema. Participants repeat the survey at 3 months post-surgery. BUE circumferential measurements are also collected before surgery and at 3 months post-surgery.
  Interventions: Other: educational intervention; Other: lymphedema survey

INTERVENTIONS:
Other: educational intervention — Receive educational handouts
  Other Names: intervention, educational
Other: lymphedema survey — Ancillary studies

SUMMARY:
This pilot clinical trial studies intensive education in increasing understanding of lymphedema in patients with breast cancer undergoing surgery. Lymphedema is the build-up of fluids in the arm (or other extremity) after surgery. Providing written educational handouts and verbal education on the risk factors and symptoms of lymphedema may improve patients' ability to identify symptoms of lymphedema after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the patient's increased knowledge of lymphedema signs/symptoms after education.

SECONDARY OBJECTIVES:

I. The participant may detect lymphedema signs/symptoms at an early stage by having a pre-surgery comparison of bilateral upper extremities (BUE) circumferential measures to the 3 month post-surgery measures.

OUTLINE:

Participants complete a five question survey, designed by the Occupational Therapy staff, as an instrument to assess a patient's knowledge of lymphedema signs/symptoms before surgery. An Occupational Therapist (OT), Physical Therapist (PT), and/or Certified Lymphedema Therapist (CLT) provide written handouts to participants on the pathophysiology, signs, symptoms, and treatment of lymphedema. Participants repeat the survey at 3 months post-surgery. BUE circumferential measurements are also collected before surgery and at 3 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be diagnosed with breast cancer; the participants will be scheduled for a lumpectomy or a mastectomy at UH GMC Seidman Cancer Center
* They must understand written, verbal, and/or recorded survey questioning English

Exclusion Criteria:

* Individuals with previous radiation treatments to the breast or axilla areas
* Prior diagnosis of lymphedema
* Persons that do not speak English
* Those unwilling to participate in the follow-up call 3 months post-surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Improvement in participant's knowledge of lymphedema | Baseline to 3 months post-surgery
  Quantitative data regarding number of correct answers to the survey questions pre-surgery and at the post-surgery 3 month re-test will be compared to assess if the lymphedema education improved the participant's knowledge of lymphedema.
Total girth differences as assessed by BUE circumferential measurements using the National Lymphedema Network (NLN) guidelines | Baseline to 3 months post-surgery
  If a > 2 cm difference is noted in girth from pre to post surgery measures, a referral will be forwarded to the physician by the study investigators and treatment options provided to the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Dotti Thompson, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States